CLINICAL TRIAL: NCT00144170
Title: Randomized, Open-label, Comparative Safety and Efficacy Study of Tipranavir Boosted With Low Dose Ritonavir (TPV/RTV) Versus Genotypically-defined Protease Inhibitor/Ritonavir (PI/RTV) in Multiple Antiretroviral Drug-experienced Patients (RESIST 2: Randomized Evaluation of Strategic Intervention in Multi-Drug Resistant Patients With Tipranavir)
Brief Title: Tipranavir/Ritonavir vs. Genotypically Defined Protease Inhibitor/Ritonavir in HIV Patients (RESIST-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1182.48; RESIST 2
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

ARMS (2):
- Tipranavir(TPV)/low dose ritonavir(r) (Other)
  Interventions: Drug: Tipranavir (with low dose ritonavir)
- Comparator protease inhibitor(CPI)/low dose ritonavir(r) (Other)
  Interventions: Drug: Comparator protease inhibitor(CPI)/low dose ritonavir(r)

INTERVENTIONS:
Drug: Tipranavir (with low dose ritonavir)
  Arms: Tipranavir(TPV)/low dose ritonavir(r)
Drug: Comparator protease inhibitor(CPI)/low dose ritonavir(r)
  Arms: Comparator protease inhibitor(CPI)/low dose ritonavir(r)

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of tipranavir/ritonavir versus an active control arm in highly treatment experienced Human immunodeficiency virus-1 infected patients. Patients must have a viral load > =1000 cells/mL, and genotype indicating at least one resistance conferring protease inhibitor-mutation as determined from a predefined panel of mutations. Any CD4+ count is acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation.
2. Human immunodeficiency virus-1 infected males or females >=18 years of age.
3. Screening genotypic resistance report indicating both of the following:

   * at least one primary protease mutation at the following sites 30N, 46I/L, 48V, 50V, 82A/F/L/T, 84V or 90M , and
   * no more than two protease mutations on codons 33, 82, 84, or 90.
4. At least 3 consecutive months experience taking antiretrovirals from each of the classes of Nucleoside reverse transcriptase inhibitor(s), Non-nucleoside reverse transcriptase inhibitor(s), and Protease inhibitor(s) at some point in treatment history,

   * with at least 2 Protease inhibitor-based regimens (minimum 3 months of exposure of each), one of which must be part of the current regimen, and
   * current Protease inhibitor-based antiretroviral medication regimen for at least 3 months prior to randomisation.
5. Human immunodeficiency virus-1 viral load >=1000 copies/mL at screening.
6. Acceptable screening laboratory values that indicate adequate baseline organ function. Laboratory values are considered to be acceptable if the following apply:

   * Total cholesterol <=400 mg/dl or 10,36 mm/L.
   * Total triglycerides <=750 mg/dl or 8,5 mm/L.
   * Alanine aminotransferase <=3x upper limit of normal and aspartate aminotransferase <=2.5x upper limit of normal.
   * Any Grade gamma-glutamyl transpeptidase is acceptable.
   * Any Grade creatinine kinase is acceptable as long as there is no concurrent myopathy.
   * All other laboratory test values <= Grade 1(Division of Acquired immune deficiency syndrome, National Institute of Health grading scale).
7. Acceptable medical history, as assessed by the investigator, with chest X-ray and electrocardiogram within 1 year of study participation.
8. Willingness to abstain from ingesting substances during the study which may alter plasma study drug levels by interaction with the cytochrome P450 system.
9. A prior Acquired immune deficiency syndrome-defining event is acceptable as long as it has resolved or the patient has been on stable treatment for at least 2 months (Acquired immune deficiency syndrome related complex is acceptable).

Exclusion Criteria:

1. Antiretroviral medication naïve.
2. Patients on recent drug holiday, defined as off antiretroviral medications for at least 7 consecutive days within the last 3 months.
3. Alanine aminotransferase >3x upper limit of normal and aspartate aminotransferase >2.5x upper limit of normal at either screening visit.
4. Female patients of child-bearing potential who:

   * have a positive serum pregnancy test at screening or during the study,
   * are breast feeding
   * are planning to become pregnant, or
   * are not willing to use a barrier method of contraception, or
   * require ethinyl estradiol administration
5. Prior tipranavir use.
6. Use of investigational medications within 30 days before study entry or during the trial. (T-20 [enfuvirtide] and Tenofovir (Viread), investigational at the time of writing of this protocol, will be allowed.)
7. Use of immunomodulatory drugs within 30 days before study entry or during the trial (e.g. interferon, cyclosporin, hydroxyurea, interleukin 2).
8. Inability to adhere to the requirements of the protocol, including active substance abuse as assessed by the investigator.
9. In the opinion of the investigator, likely survival of less than 12 months because of underlying disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2003-02; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (174):
- Argentina (6):
  - 1182.48.5401 Fundación Huésped, Buenos Aires
  - 1182.48.5402 Fundación Huésped, Buenos Aires
  - 1182.48.5403 Servicio de Infecciosas, Buenos Aires
  - 1182.48.5404 Servicio de Infecciosas, Buenos Aires
  - 1182.48.5405 Hospital Muniz, Buenos Aires
  - 1182.48.5406 Servicio de Immunocomprometido, Buenos Aires
- 1182.48.4301 Boehringer Ingelheim Investigational Site, Vienna, Austria
- Belgium (6):
  - 1182.48.3209 Boehringer Ingelheim Investigational Site, Antwerp
  - 1182.48.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.48.3202 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.48.3206 Boehringer Ingelheim Investigational Site, Charleroi
  - 1182.48.3207 Boehringer Ingelheim Investigational Site, Ghent
  - 1182.48.3210 Boehringer Ingelheim Investigational Site, Luxembourg
- Brazil (13):
  - 1182.48.5512 Cidade Universitária Zeferino Vaz-Clínica Médica FCM, Campinas - SP
  - 1182.48.5505 Instituto A-Z de Pesquisa e Ensino da PUC, Curitiba - PR
  - 1182.48.5507 Hospital Geral de Nova Iguaçu - Ministério da Saúde, Nova Iguaçu - RJ
  - 1182.48.5502 Fundação Oswaldo Cruz, Rio de Janeiro - RJ
  - 1182.48.5509 Universidade Federal do Rio de Janeiro, Rio de Janeiro - RJ
  - 1182.48.5511 Universidade Federal da Bahia-Unidade Docente Assistencial d, Salvador - BA
  - 1182.48.5501 Clínica de Doenças Parasitárias e Infecciosas-Hospital Dia, São Paulo - SP
  - 1182.48.5503 I.I. Emilio Ribas - Moléstias Infecciosas, São Paulo - SP
  - 1182.48.5504 Hospital do Servidor Público Estadual - IAMSPE, São Paulo - SP
  - 1182.48.5506 Centro de Referência e Treinamento - DST/AIDS, São Paulo - SP
  - 1182.48.5508 I.I. Emilio Ribas, São Paulo - SP
  - 1182.48.5510 INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo - SP
  - 1182.48.5513 UNIFESP - Centro de Pesquisa Clinica, São Paulo - SP
- Denmark (4):
  - 1182.48.4505 Boehringer Ingelheim Investigational Site, Aarhus N
  - 1182.48.4502 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1182.48.4501 Boehringer Ingelheim Investigational Site, København Ø
  - 1182.48.4504 Boehringer Ingelheim Investigational Site, Odense C
- France (23):
  - 1182.48.3311 Boehringer Ingelheim Investigational Site, Besançon
  - 1182.48.3307 Boehringer Ingelheim Investigational Site, Bordeaux
  - 1182.48.3317 Boehringer Ingelheim Investigational Site, Bordeaux
  - 1182.48.3302 Boehringer Ingelheim Investigational Site, Caen
  - 1182.48.3303 Boehringer Ingelheim Investigational Site, Clamart
  - 1182.48.3305 Boehringer Ingelheim Investigational Site, Le Kremlin-Bicêtre
  - 1182.48.3304 Boehringer Ingelheim Investigational Site, Lyon
  - 1182.48.3322 Boehringer Ingelheim Investigational Site, Lyon
  - 1182.48.3308 Boehringer Ingelheim Investigational Site, Marseille
  - 1182.48.3309 Boehringer Ingelheim Investigational Site, Marseille
  - 1182.48.3318 Boehringer Ingelheim Investigational Site, Nantes
  - 1182.48.3306 Boehringer Ingelheim Investigational Site, Nice
  - 1182.48.3301 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3310 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3312 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3316 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3319 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3321 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3323 Boehringer Ingelheim Investigational Site, Paris
  - 1182.48.3315 Boehringer Ingelheim Investigational Site, Rennes
  - 1182.48.3313 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1182.48.3314 Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
  - 1182.48.3320 Boehringer Ingelheim Investigational Site, Villejuif
- Germany (28):
  - 1182.48.4911 Boehringer Ingelheim Investigational Site, Aachen
  - 1182.48.4901 Boehringer Ingelheim Investigational Site, Berlin
  - 1182.48.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1182.48.4903 Boehringer Ingelheim Investigational Site, Bochum
  - 1182.48.4918 Boehringer Ingelheim Investigational Site, Bonn
  - 1182.48.4905 Boehringer Ingelheim Investigational Site, Cologne
  - 1182.48.4926 Boehringer Ingelheim Investigational Site, Cologne
  - 1182.48.4906 Boehringer Ingelheim Investigational Site, Dortmund
  - 1182.48.4912 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1182.48.4914 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1182.48.4908 Boehringer Ingelheim Investigational Site, Erlangen
  - 1182.48.4904 Boehringer Ingelheim Investigational Site, Essen
  - 1182.48.4924 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1182.48.4928 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1182.48.4930 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1182.48.4916 Boehringer Ingelheim Investigational Site, Hamburg
  - 1182.48.4929 Boehringer Ingelheim Investigational Site, Hamburg
  - 1182.48.4931 Boehringer Ingelheim Investigational Site, Hamburg
  - 1182.48.4913 Boehringer Ingelheim Investigational Site, Hanover
  - 1182.48.4920 Boehringer Ingelheim Investigational Site, Hanover
  - 1182.48.4909 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1182.48.4923 Boehringer Ingelheim Investigational Site, Mannheim
  - 1182.48.4907 Boehringer Ingelheim Investigational Site, München
  - 1182.48.4910 Boehringer Ingelheim Investigational Site, München
  - 1182.48.4915 Boehringer Ingelheim Investigational Site, Osnabrück
  - 1182.48.4919 Boehringer Ingelheim Investigational Site, Regensburg
  - 1182.48.4921 Boehringer Ingelheim Investigational Site, Stuttgart
  - 1182.48.4927 Boehringer Ingelheim Investigational Site, Stuttgart
- Greece (10):
  - 1182.48.3001 Boehringer Ingelheim Investigational Site, Athens
  - 1182.48.3002 Boehringer Ingelheim Investigational Site, Athens
  - 1182.48.3003 Boehringer Ingelheim Investigational Site, Athens
  - 1182.48.3004 Boehringer Ingelheim Investigational Site, Athens
  - 1182.48.3006 Boehringer Ingelheim Investigational Site, Athens
  - 1182.48.3007 Boehringer Ingelheim Investigational Site, Athens
  - 1182.48.3005 Boehringer Ingelheim Investigational Site, Goudi, Athens
  - 1182.48.3010 Boehringer Ingelheim Investigational Site, Pátrai
  - 1182.48.3008 Boehringer Ingelheim Investigational Site, Peraeus
  - 1182.48.3009 Boehringer Ingelheim Investigational Site, Thessaloniki
- 1182.48.3531 Boehringer Ingelheim Investigational Site, Dublin, Ireland
- Italy (30):
  - 1182.48.3930 Boehringer Ingelheim Investigational Site, Ancona
  - 1182.48.3920 Boehringer Ingelheim Investigational Site, Antella (fi)
  - 1182.48.3926 Boehringer Ingelheim Investigational Site, Bari
  - 1182.48.3932 Boehringer Ingelheim Investigational Site, Bergamo
  - 1182.48.3908 Boehringer Ingelheim Investigational Site, Brescia
  - 1182.48.3929 Boehringer Ingelheim Investigational Site, Busto Arsizio (va)
  - 1182.48.3917 Boehringer Ingelheim Investigational Site, Ferrara
  - 1182.48.3919 Boehringer Ingelheim Investigational Site, Florence
  - 1182.48.3905 Boehringer Ingelheim Investigational Site, Genova
  - 1182.48.3927 Boehringer Ingelheim Investigational Site, Genova
  - 1182.48.3925 Boehringer Ingelheim Investigational Site, Lecco
  - 1182.48.3910 Boehringer Ingelheim Investigational Site, Macerata
  - 1182.48.3901 Boehringer Ingelheim Investigational Site, Milan
  - 1182.48.3907 Boehringer Ingelheim Investigational Site, Milan
  - 1182.48.3924 Boehringer Ingelheim Investigational Site, Milan
  - 1182.48.3934 Boehringer Ingelheim Investigational Site, Milan
  - 1182.48.3915 Boehringer Ingelheim Investigational Site, Modena
  - 1182.48.3912 Boehringer Ingelheim Investigational Site, Napoli
  - 1182.48.3921 Boehringer Ingelheim Investigational Site, Padua
  - 1182.48.3916 Boehringer Ingelheim Investigational Site, Pavia
  - 1182.48.3922 Boehringer Ingelheim Investigational Site, Pavia
  - 1182.48.3904 Boehringer Ingelheim Investigational Site, Rimini
  - 1182.48.3902 Boehringer Ingelheim Investigational Site, Roma
  - 1182.48.3903 Boehringer Ingelheim Investigational Site, Roma
  - 1182.48.3909 Boehringer Ingelheim Investigational Site, Roma
  - 1182.48.3935 Boehringer Ingelheim Investigational Site, Roma
  - 1182.48.3906 Boehringer Ingelheim Investigational Site, Torino
  - 1182.48.3914 Boehringer Ingelheim Investigational Site, Torino
  - 1182.48.3931 Boehringer Ingelheim Investigational Site, Torino
  - 1182.48.3933 Boehringer Ingelheim Investigational Site, Treviso
- Mexico (4):
  - 1182.48.5201 Centro Médico La Raza IMSS, Mexico City
  - 1182.48.5202 Hospital Lopez Mateos, México
  - 1182.48.5203 Centro Guadalajara, Jal., México
  - 1182.48.5206 Centro Medico San Vicente, Monterrey, N.l.
- Netherlands (6):
  - 1182.48.3101 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1182.48.3106 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1182.48.3108 Boehringer Ingelheim Investigational Site, Groningen
  - 1182.48.3105 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1182.48.3104 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1182.48.3110 Boehringer Ingelheim Investigational Site, The Hague
- Portugal (5):
  - 1182.48.3502 Boehringer Ingelheim Investigational Site, Cascais
  - 1182.48.3503 Boehringer Ingelheim Investigational Site, Coimbra
  - 1182.48.3501 Boehringer Ingelheim Investigational Site, Lisbon
  - 1182.48.3505 Hospital Egas Moniz, Lisbon
  - 1182.48.3504 Hospital de São João, Porto
- Spain (19):
  - 1182.48.3415 Boehringer Ingelheim Investigational Site, Alicante
  - 1182.48.3405 Boehringer Ingelheim Investigational Site, Badalona
  - 1182.48.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.48.3407 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.48.3408 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.48.3409 Boehringer Ingelheim Investigational Site, Barcelona
  - 1182.48.3416 Boehringer Ingelheim Investigational Site, Donostia / San Sebastian
  - 1182.48.3406 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1182.48.3402 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.48.3403 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.48.3404 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.48.3410 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.48.3411 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.48.3412 Boehringer Ingelheim Investigational Site, Madrid
  - 1182.48.3417 Boehringer Ingelheim Investigational Site, Málaga
  - 1182.48.3413 Boehringer Ingelheim Investigational Site, Seville
  - 1182.48.3414 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.48.3420 Boehringer Ingelheim Investigational Site, Valencia
  - 1182.48.3418 Boehringer Ingelheim Investigational Site, Vigo
- Sweden (3):
  - 1182.48.4603 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1182.48.4602 Boehringer Ingelheim Investigational Site, Malmo
  - 1182.48.4601 Boehringer Ingelheim Investigational Site, Stockholm
- Switzerland (4):
  - 1182.48.4101 Universitätsspital Basel, Basel
  - 1182.48.4104 Hopital Universitaire de Genève, Geneva
  - 1182.48.4103 Kantonsspital St. Gallen, Sankt Gallen
  - 1182.48.4102 Universitätsspital Zürich, Zurich
- United Kingdom (11):
  - 1182.48.4405 Boehringer Ingelheim Investigational Site, Brighton
  - 1182.48.4412 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1182.48.4411 Boehringer Ingelheim Investigational Site, Liverpool
  - 1182.48.4404 Boehringer Ingelheim Investigational Site, London
  - 1182.48.4406 Boehringer Ingelheim Investigational Site, London
  - 1182.48.4408 Boehringer Ingelheim Investigational Site, London
  - 1182.48.4409 Boehringer Ingelheim Investigational Site, London
  - 1182.48.4414 Boehringer Ingelheim Investigational Site, London
  - 1182.48.4418 Boehringer Ingelheim Investigational Site, London
  - 1182.48.4417 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1182.48.4407 Boehringer Ingelheim Investigational Site, Portsmouth

REFERENCES:
- [Derived] Mikl J, Sulkowski MS, Benhamou Y, Dieterich D, Pol S, Rockstroh J, Robinson PA, Ranga M, Stern JO. Hepatic profile analyses of tipranavir in Phase II and III clinical trials. BMC Infect Dis. 2009 Dec 14;9:203. doi: 10.1186/1471-2334-9-203. PMID 20003457
- [Derived] Hicks CB, Cahn P, Cooper DA, Walmsley SL, Katlama C, Clotet B, Lazzarin A, Johnson MA, Neubacher D, Mayers D, Valdez H; RESIST investigator group. Durable efficacy of tipranavir-ritonavir in combination with an optimised background regimen of antiretroviral drugs for treatment-experienced HIV-1-infected patients at 48 weeks in the Randomized Evaluation of Strategic Intervention in multi-drug reSistant patients with Tipranavir (RESIST) studies: an analysis of combined data from two randomised open-label trials. Lancet. 2006 Aug 5;368(9534):466-75. doi: 10.1016/S0140-6736(06)69154-X. PMID 16890833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The discrepancy with enrollment number in the protocol section is due to 16 patients not treated. (7 from TPV/r and 9 from CPI/r). These patients were not included in any analyses or results.
Period: Overall Study
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Started | 438 | 428
Completed | 86 | 32
Not Completed | 352 | 396
Not completed — Adverse Event | 84 | 41
Not completed — Protocol Violation | 23 | 16
Not completed — Lost to Follow-up | 5 | 10
Not completed — Withdrawal by Subject | 29 | 13
Not completed — Other reason not defined above | 211 | 316

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPI)/Low Dose Ritonavir(r) | Total
Number analyzed (Participants) | 435 | 428 | 863
Age, Continuous [Mean (Standard Deviation); unit: years] — 3 patients were not randomized but treated with TPV/r. They are included in the participant flow and adverse events but not in the efficacy analysis.
  years | 42.5 (8.4) | 42.9 (8) | 42.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — 3 patients were not randomized but treated with TPV/r. They are included in the participant flow and adverse events but not in the efficacy analysis.
  Participants
    Female | 84 | 64 | 148
    Male | 351 | 364 | 715

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response at Week 48
Description: Patients who experienced treatment response. Treatment response (TR) is defined as two consecutive VL ≥ 1 log10 below baseline without discontinuation of study drug, change in anti-retroviral background, or rebound
Time Frame: after 48 weeks of treatment
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 34.5 | 15
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 18.5, 95% CI 2-sided [12.9 to 24.0]

2. Primary Outcome: Time to Treatment Failure Through 48 Weeks of Treatment
Description: Time to treatment failure is defined as 0 for patients who never achieve TR otherwise time to treatment failure is the earliest time of death, discontinuation of the study drug or introduction of a new anti-retroviral drug to the regimen if it is not solely related to either toxicity or intolerance clearly attributable to a background, or the first of two consecutive visits with Log(baseline Viral Load) - Log(on-treatment Viral Load) < 1.
Time Frame: after 48 weeks of treatment
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Days | 112 [0 to 475] | 0 [0 to 112]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

3. Secondary Outcome: Treatment Response at Week 2
Description: as for outcome 1
Time Frame: week 2
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 51 | 25.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 24.9, 95% CI 2-sided [18.6 to 31.1]

4. Secondary Outcome: Treatment Response at Week 4
Description: as for outcome 1
Time Frame: week 4
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 59.1 | 29.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.8, 95% CI 2-sided [22.5 to 35.1]

5. Secondary Outcome: Treatment Response at Week 8
Description: as for outcome 1
Time Frame: week 8
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 54.3 | 24.5
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 29.4, 95% CI 2-sided [23.2 to 35.7]

6. Secondary Outcome: Treatment Response at Week 16
Description: as for outcome 1
Time Frame: week 16
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 47.1 | 19.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 26.6, 95% CI 2-sided [20.5 to 32.6]

7. Secondary Outcome: Treatment Response at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 40.9 | 18.0
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 22.1, 95% CI 2-sided [16.2 to 27.9]

8. Secondary Outcome: Treatment Response at Week 32
Description: as for outcome 1
Time Frame: week 32
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 37.2 | 17.3
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 19.0, 95% CI 2-sided [13.3 to 24.7]

9. Secondary Outcome: Treatment Response at Week 40
Description: as for outcome 1
Time Frame: week 40
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 36.3 | 16.6
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 18.7, 95% CI 2-sided [13.0 to 24.4]

10. Secondary Outcome: Treatment Response at Week 56
Description: as for outcome 1
Time Frame: week 56
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 32.6 | 14.5
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 17.2, 95% CI 2-sided [11.7 to 22.7]

11. Secondary Outcome: Treatment Response at Week 64
Description: as for outcome 1
Time Frame: week 64
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 31 | 13.3
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 17.1, 95% CI 2-sided [11.7 to 22.4]

12. Secondary Outcome: Treatment Response at Week 72
Description: as for outcome 1
Time Frame: week 72
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 30.1 | 12.1
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 17.3, 95% CI 2-sided [12.0 to 22.5]

13. Secondary Outcome: Treatment Response at Week 80
Description: as for outcome 1
Time Frame: week 80
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 28.5 | 11.4
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 16.4, 95% CI 2-sided [11.2 to 21.5]

14. Secondary Outcome: Treatment Response at Week 88
Description: as for outcome 1
Time Frame: week 88
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 27.8 | 11
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 16.2, 95% CI 2-sided [11.1 to 21.3]

15. Secondary Outcome: Treatment Response at Week 96
Description: as for outcome 1
Time Frame: after 96 weeks of treatment
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
percentage of participants | 26.2 | 10
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Weighted by the size of enfuvirtide and protease inhibitor strata; Risk Difference (RD) = 15.6, 95% CI 2-sided [10.6 to 20.6]

16. Secondary Outcome: Time to Treatment Failure Through 96 Weeks of Treatment
Description: as for outcome 2
Time Frame: after 96 weeks of treatment
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Days | 115 [0 to 811] | 0 [0 to 112]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

17. Secondary Outcome: Time to Confirmed Virologic Failure Through 48 Weeks of Treatment
Description: Time to virologic failure is defined as the time from the start of treatment to the last measurement where the Log(baseline viral load)-Log(on-treatment viral load)>1 before a 2 consecutive measurements where Log(baseline viral load)-Log(on-treatment viral load)<1.
Time Frame: after 48 weeks of treatment
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Days | 117 [0 to 475] | 0 [0 to 112]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

18. Secondary Outcome: Time to Confirmed Virologic Failure Through 96 Weeks of Treatment
Description: as for outcome 17
Time Frame: after 96 weeks of treatment
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Days | 117 [0 to 756] | 0 [0 to 112]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

19. Secondary Outcome: Virologic Response
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: Week 2 through Week 96 (at any point during trial)
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 75.6 | 48.6

20. Secondary Outcome: Virologic Response at Week 2
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: Week 2
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 60.5 | 36

21. Secondary Outcome: Virologic Response at Week 4
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 4
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 62.3 | 33.4

22. Secondary Outcome: Virologic Response at Week 8
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 8
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 56.3 | 26.6

23. Secondary Outcome: Virologic Response at Week 16
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 16
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 47.1 | 20.8

24. Secondary Outcome: Virologic Response at Week 24
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 24
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 42.8 | 19.2

25. Secondary Outcome: Virologic Response at Week 32
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 32
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 38.6 | 19.4

26. Secondary Outcome: Virologic Response at Week 40
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 40
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 37 | 17.3

27. Secondary Outcome: Virologic Response at Week 48
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 48
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 36.8 | 16.6

28. Secondary Outcome: Virologic Response at Week 56
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 56
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 35.2 | 15.2

29. Secondary Outcome: Virologic Response at Week 64
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: week 64
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 33.6 | 14

30. Secondary Outcome: Virologic Response at Week 72
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: Week 72
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 32.2 | 13.8

31. Secondary Outcome: Virologic Response at Week 80
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: Week 80
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 32.6 | 13.6

32. Secondary Outcome: Virologic Response at Week 88
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: Week 88
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 31 | 12.1

33. Secondary Outcome: Virologic Response at Week 96
Description: Virologic response is defined as: Log(baseline viral load (VL))-Log(on-treatment VL)>=1
Time Frame: Week 96
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 30.1 | 11.4

34. Secondary Outcome: Median Change From Baseline in Viral Load (Week 2)
Time Frame: Baseline to Week 2
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -1.27 [-1.78 to -0.55] | -0.56 [-1.28 to 0]

35. Secondary Outcome: Median Change From Baseline in Viral Load (Week 4)
Time Frame: Baseline to Week 4
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -1.47 [-2.03 to -0.4] | -0.42 [-1.35 to 0]

36. Secondary Outcome: Median Change From Baseline in Viral Load (Week 8)
Time Frame: Baseline to Week 8
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -1.4 [-2.25 to -0.22] | -0.33 [-1.23 to 0]

37. Secondary Outcome: Median Change From Baseline in Viral Load (Week 16)
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -1.03 [-2.35 to -0.17] | -0.3 [-0.93 to -0.02]

38. Secondary Outcome: Median Change From Baseline in Viral Load (Week 24)
Time Frame: Baseline to Week 24
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.69 [-2.28 to -0.11] | -0.21 [-0.86 to 0.06]

39. Secondary Outcome: Median Change From Baseline in Viral Load (Week 32)
Time Frame: Baseline to Week 32
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.63 [-2.29 to -0.09] | -0.24 [-0.84 to 0.06]

40. Secondary Outcome: Median Change From Baseline in Viral Load (Week 40)
Time Frame: Baseline to Week 40
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.65 [-2.27 to -0.07] | -0.2 [-0.73 to 0.1]

41. Secondary Outcome: Median Change From Baseline in Viral Load (Week 48)
Time Frame: Baseline to Week 48
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.65 [-2.17 to -0.07] | -0.2 [-0.75 to 0.11]

42. Secondary Outcome: Median Change From Baseline in Viral Load (Week 56)
Time Frame: Baseline to Week 56
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.64 [-2.16 to -0.07] | -0.22 [-0.74 to 0.11]

43. Secondary Outcome: Median Change From Baseline in Viral Load (Week 64)
Time Frame: Baseline to Week 64
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.63 [-2.12 to -0.07] | -0.21 [-0.71 to 0.12]

44. Secondary Outcome: Median Change From Baseline in Viral Load (Week 72)
Time Frame: Baseline to Week 72
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.52 [-2.14 to -0.05] | -0.2 [-0.7 to 0.11]

45. Secondary Outcome: Median Change From Baseline in Viral Load (Week 80)
Time Frame: Baseline to Week 80
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.55 [-2.14 to -0.06] | -0.2 [-0.72 to 0.11]

46. Secondary Outcome: Median Change From Baseline in Viral Load (Week 88)
Time Frame: Baseline to Week 88
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.56 [-2.12 to -0.03] | -0.2 [-0.7 to 0.11]

47. Secondary Outcome: Median Change From Baseline in Viral Load (Week 96)
Time Frame: Baseline to Week 96
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Log(Copies/mL) | -0.56 [-2.14 to -0.05] | -0.2 [-0.67 to 0.11]

48. Secondary Outcome: Virologic Response at Week 40
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 40
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 31.5 | 15

49. Secondary Outcome: Virologic Response at Viral Load Nadir During Study Treatment Through 96 Weeks
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 2 through Week 96 (at any point during trial)
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 52.2 | 25.7

50. Secondary Outcome: Virologic Response at Week 2
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 2
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 14.5 | 8.2

51. Secondary Outcome: Virologic Response at Week 4
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 4
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 26.2 | 15.2

52. Secondary Outcome: Virologic Response at Week 8
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 8
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 33.3 | 17.5

53. Secondary Outcome: Virologic Response at Week 16
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 16
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 35.2 | 17.5

54. Secondary Outcome: Virologic Response at Week 24
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 24
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 32.6 | 15.4

55. Secondary Outcome: Virologic Response at Week 32
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 32
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 32.4 | 16.1

56. Secondary Outcome: Virologic Response at Week 48
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 48
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 30.1 | 13.6

57. Secondary Outcome: Virologic Response at Week 56
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 56
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 30.6 | 12.4

58. Secondary Outcome: Virologic Response at Week 64
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 64
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 28.7 | 12.1

59. Secondary Outcome: Virologic Response at Week 72
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 72
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 28 | 11.4

60. Secondary Outcome: Virologic Response at Week 80
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: Week 80
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 28.7 | 11

61. Secondary Outcome: Virologic Response at Week 88
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: week 88
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 27.8 | 11.2

62. Secondary Outcome: Virologic Response at Week 96
Description: Virologic response defined as Viral Load<400 copies/mL
Time Frame: week 96
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 27.1 | 10.3

63. Secondary Outcome: Virologic Response
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 2 through Week 96 (at any point during trial)
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 36.6 | 16.8

64. Secondary Outcome: Virologic Response at Week 2
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 2
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 0.9 | 1.4

65. Secondary Outcome: Virologic Response at Week 4
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 4
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 4.4 | 3.5

66. Secondary Outcome: Virologic Response at Week 8
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 8
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 11 | 6.8

67. Secondary Outcome: Virologic Response at Week 16
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 16
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 20.5 | 10.5

68. Secondary Outcome: Virologic Response at Week 24
Description: Viral Load < 50 copies/mL
Time Frame: Week 24
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 21.1 | 11.9

69. Secondary Outcome: Virologic Response at Week 32
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 32
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 22.1 | 12.1

70. Secondary Outcome: Virologic Response at Week 40
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 40
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 22.3 | 11.9

71. Secondary Outcome: Virologic Response at Week 48
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 48
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 22.8 | 10.5

72. Secondary Outcome: Virologic Response at Week 56
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 56
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 22.5 | 8.9

73. Secondary Outcome: Virologic Response at Week 64
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 64
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 21.6 | 8.2

74. Secondary Outcome: Virologic Response at Week 72
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 72
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 21.1 | 8.2

75. Secondary Outcome: Virologic Response at Week 80
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 80
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 21.8 | 8.9

76. Secondary Outcome: Virologic Response at Week 88
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 88
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 20.7 | 8.9

77. Secondary Outcome: Virologic Response at Week 96
Description: Virologic response defined as Viral Load<50 copies/mL
Time Frame: Week 96
Population: Full Analysis Set (FAS), included all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Percentage of participants | 20 | 8.9

78. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 2)
Time Frame: Baseline to Week 2
Population: Full Analysis Set having baseline CD4 (FAS CD4), included all randomized patients treated with at least one dose of study medication having baseline CD4 count
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 26 (65) | 13 (56)

79. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 4)
Time Frame: Baseline to Week 4
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 39 (77) | 19 (64)

80. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 8)
Time Frame: Baseline to Week 8
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 52 (85) | 25 (76)

81. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 16)
Time Frame: Baseline to Week 16
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 57 (90) | 25 (77)

82. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 24)
Time Frame: Baseline to Week 24
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 51 (97) | 21 (81)

83. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 32)
Time Frame: Baseline to Week 32
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 46 (102) | 17 (87)

84. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 40)
Time Frame: Baseline to Week 40
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 47 (99) | 19 (87)

85. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 48)
Time Frame: Baseline to Week 48
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 43 (109) | 16 (92)

86. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 56)
Time Frame: Baseline to Week 56
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 39 (113) | 16 (95)

87. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 64)
Time Frame: Baseline to Week 64
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 42 (125) | 13 (92)

88. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 72)
Time Frame: Baseline to Week 72
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 42 (129) | 18 (105)

89. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 80)
Time Frame: Baseline to Week 80
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 39 (125) | 19 (112)

90. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 88)
Time Frame: Baseline to Week 88
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 41 (138) | 19 (109)

91. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count (Week 96)
Time Frame: Baseline to Week 96
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 430 | 418
Cells/mm3 | 41 (132) | 20 (111)

92. Secondary Outcome: Time to New Centers for Disease Control (CDC) Class C Progression Event or Death.
Description: Time to death or occurrence of AIDS-defining condition according to the US Centers for Disease Control and Prevention case definition.
  The median and quartiles are underestimated since more than 92% of the observations (in both treatment arms) were censored and the estimation was restricted to the largest observed event time.
Time Frame: up to 75 weeks of treatment
Population: Safety Set (SAF), included all patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 435 | 428
Days | 528 [528 to 528] | 332 [332 to 332]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparator Protease Inhibitor(CPI)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.1026, Log Rank

ADVERSE EVENTS:
Time Frame: 240 weeks
Description: 3 patients were not randomized but treated with TPV/r. They are included in the participant flow and adverse events but not in the efficacy analysis.
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPI)/Low Dose Ritonavir(r)
Serious Adverse Events (participants affected / at risk) | 123/438 | 89/428
Other Adverse Events (participants affected / at risk) | 359/438 | 270/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir(TPV)/Low Dose Ritonavir(r) (N=438) | Comparitor Protease Inhibitor(CPI)/Low Dose Ritonavir(r) (N=428)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Chorioretinitis (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 1
Retinitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 5 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 2 | 2
Local swelling (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 13 | 9
Sudden death (General disorders) | 0 | 1
Cholangitis chronic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
AIDS encephalopathy (Infections and infestations) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Actinomycotic pulmonary infection (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 2
Anal infection (Infections and infestations) | 1 | 0
Anogenital warts (Infections and infestations) | 4 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Campylobacter intestinal infection (Infections and infestations) | 1 | 0
Cerebral toxoplasmosis (Infections and infestations) | 3 | 4
Cryptosporidiosis infection (Infections and infestations) | 0 | 1
Cyclosporidium infection (Infections and infestations) | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 2 | 3
Cytomegalovirus colitis (Infections and infestations) | 2 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 2 | 0
Disseminated cryptococcosis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 4
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
HIV infection (Infections and infestations) | 1 | 0
Haemophilus sepsis (Infections and infestations) | 0 | 1
Helicobacter sepsis (Infections and infestations) | 1 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Histoplasmosis (Infections and infestations) | 0 | 1
Isosporiasis (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 3 | 3
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 1
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 11 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 2 | 3
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Salmonella sepsis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0
Syphilis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 0 | 1
Visceral leishmaniasis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Accident at home (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood lactic acid increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Electrocardiogram change (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 3 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Mitochondrial toxicity (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hodgkin's disease mixed cellularity stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral ataxia (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical root pain (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 3
Hemiparesis (Nervous system disorders) | 2 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 2
Lacunar infarction (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 2
Depression suicidal (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrogenic diabetes insipidus (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Eventration procedure (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir(TPV)/Low Dose Ritonavir(r) (N=438) | Comparitor Protease Inhibitor(CPI)/Low Dose Ritonavir(r) (N=428)
Abdominal pain (Gastrointestinal disorders) | 50 | 29
Abdominal pain upper (Gastrointestinal disorders) | 35 | 25
Diarrhoea (Gastrointestinal disorders) | 148 | 100
Dyspepsia (Gastrointestinal disorders) | 27 | 18
Flatulence (Gastrointestinal disorders) | 27 | 18
Nausea (Gastrointestinal disorders) | 87 | 42
Vomiting (Gastrointestinal disorders) | 57 | 34
Adverse drug reaction (General disorders) | 22 | 2
Asthenia (General disorders) | 34 | 26
Fatigue (General disorders) | 39 | 24
Pyrexia (General disorders) | 65 | 39
Bronchitis (Infections and infestations) | 58 | 23
Influenza (Infections and infestations) | 48 | 35
Nasopharyngitis (Infections and infestations) | 74 | 38
Oral candidiasis (Infections and infestations) | 42 | 31
Sinusitis (Infections and infestations) | 36 | 16
Urinary tract infection (Infections and infestations) | 26 | 6
Weight decreased (Investigations) | 32 | 14
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 32 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 13
Dizziness (Nervous system disorders) | 39 | 15
Headache (Nervous system disorders) | 78 | 34
Depression (Psychiatric disorders) | 31 | 14
Insomnia (Psychiatric disorders) | 27 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 16
Rash (Skin and subcutaneous tissue disorders) | 36 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.